CLINICAL TRIAL: NCT02969148
Title: Laparoscopic Bursectomy and D2 Lymphadenectomy vs.Laparoscopic D2 Lymphadenectomy in II,III Stage Gastric Carcinoma: A Prospective, Randomized, Single Blind, Parallel Group Clinical Trial
Brief Title: Laparoscopic Bursectomy and D2 Lymphadenectomy vs.Laparoscopic D2 Lymphadenectomy in Advanced Gastric Cancer
Acronym: LBDL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Jin Wan, professor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LBDL1
Record Dates: First submitted 2016-11-10; First posted 2016-11-21 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Gastric Cancer Stage II; Gastric Cancer Stage III
Keywords: Laparoscopic; Bursectomy; D2 lymphadenectomy; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The bursectomy and D2 lymphadenectomy (Experimental): Laparoscopic bursectomy and D2 lymphadenectomy will be performed for the treatment of patients assigned to this group.The key of this approach are that anterior lobe of transverse mesocolon and capsula pancreatis will be dissected with the D2 lymphadenectomy according to the guidelines of National Comprehensive Cancer Network(NCCN)
  Interventions: Procedure: Laparoscopic bursectomy and D2 lymphadenectomy
- The D2 lymphadenectomy (Active Comparator): Laparoscopic D2 lymphadenectomy will be performed for the treatment of patients assigned to this group.The key of this approach is that D2 lymphadenectomy is carried out according to the guidelines of National Comprehensive Cancer Network(NCCN) without dissociation of anterior lobe of transverse mesocolon and capsula pancreatis.
  Interventions: Procedure: Laparoscopic D2 lymphadenectomy

INTERVENTIONS:
Procedure: Laparoscopic bursectomy and D2 lymphadenectomy — The anterior lobe of transverse mesocolon and capsula pancreatis will be dissected with the D2 lymphadenectomy according to the guidelines of National Comprehensive Cancer Network(NCCN) by laparoscopy，this is Laparoscopic bursectomy and D2 lymphadenectomy.
  Arms: The bursectomy and D2 lymphadenectomy
Procedure: Laparoscopic D2 lymphadenectomy — D2 lymphadenectomy is carried out according to the guidelines of National Comprehensive Cancer Network(NCCN).
  Arms: The D2 lymphadenectomy

SUMMARY:
To investigate the clinical efficacy and safety of laparoscopic bursectomy and D2 lymphadenectomy (LBDL group) versus laparoscopic D2 lymphadenectomy (LDL group) in advanced gastric cancer by prospective randomized controlled clinical trial.

DETAILED DESCRIPTION:
To compare the LBDL group and LDL group in the advanced gastric cancer. A prospective randomized controlled trial will be performed in the GI department, Guangdong provincial hospital of Chinese Medicine from November 2016 to November 2024. The sample size，100 cases with advanced gastric cancer, will be needed after calculated by the statistics. The 100 cases will be randomly divided into two groups: LBDL group and LDL group. Primary outcomes are the 3 years' Disease-free survival (DFS) rate, The secondary outcomes are the 3 years' and 5 years' Disease-free survival (DFS) rate, the 3 years and 5 years Overall survival（OS）rate, operative time, the total blood loss, the intra-operative complication and the post-operative complication, the number of lymph nodes dissected, the number of conversion to open laparotomy, and the other outcomes are the average time of ground activities, the hospital stay. The data in two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. The age limits is 18-80 years old;
2. T3-T4 resectable gastric carcinoma,confirmed by CT and pathology.
3. The preoperative imaging confirmed that the tumor did not involve adjacent organs;
4. American Society of anesthesiologists (ASA) score less than or equal to Level 3;
5. Criteria of performance status karnofsky is greater than or equal to 60.

Exclusion Criteria:

1. The patients' age limits is Less than 18 years old, or more than 80 years old;
2. The preoperative imaging confirmed that the tumor involve adjacent organs;
3. The tumor have been finding distant metastases;
4. American Society of anesthesiologists (ASA) score more than 3;
5. Criteria of performance status karnofsky is lower than 60;
6. There is a laparoscopic surgery contraindications.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2022-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
the 3-year disease-free survival rate | up to 36 months

SECONDARY OUTCOMES:
the 3-year overall survival rate | up to 36 months
the 5-year disease-free survival rate | up to 5 years
the 5-year overall survival rate | up to 5 years
the operation time | up to 36 months
the total blood loss | up to 36 months
the number of pancreatic leakage | up to 36 months
the number of lymph nodes dissected | up to 36 months
the number of conversion to open laparotomy | up to 36 months
the number of bowel obstruction | up to 36 months

OTHER OUTCOMES:
the time to firstly flaunt | up to 36 months
the time of hospital stay | up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Jin Wan, professor, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine; Liao-nan Zou, professor, Study Director — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- GI surgery,Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Zou LN, He YB, Li HM, Diao DC, Mo DL, Wang W, Wan J. Surgical skills for laparoscopic resection of the bursa omentalis and lymph node scavenging with radical gastrectomy. Oncol Lett. 2015 Jul;10(1):99-102. doi: 10.3892/ol.2015.3226. Epub 2015 May 19. PMID 26170983
- [Result] Zou L, Xiong W, Mo D, Chen G, He Y, Li H, Tan P, Wang W, Wan J. Totally laparoscopic complete bursectomy and D2 lymphadenectomy in radical total gastrectomy: an outside bursa omentalis approach. Surg Endosc. 2016 Sep;30(9):4152. doi: 10.1007/s00464-015-4702-z. Epub 2015 Dec 16. PMID 26675932